CLINICAL TRIAL: NCT05292976
Title: Multi-center, Randomized, Double Blind, Double Dummy, Placebo and Active Controlled, Crossover Pharmacodynamic Bioequivalence Study of Albuterol Sulfate Inhalation Aerosol, 0.09 mg in Stable Mild Asthma Patients
Brief Title: Pharmacodynamic Bioequivalence Study of Albuterol Sulfate Inhalation Aerosol, 0.09 mg Albuterol Base/ Inhalation
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Aurobindo Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR206-19
Record Dates: First submitted 2022-03-15; First posted 2022-03-23 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Dummy
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Zero dose: (Placebo Comparator)
  Interventions: Other: Methacholine Chloride; Drug: Placebo
- Reference 0.09 mg (Active Comparator)
  Interventions: Other: Methacholine Chloride; Drug: Albuterol Sulfate HFA 0.09 mg (Reference)
- Reference 0.18 mg (Active Comparator)
  Interventions: Other: Methacholine Chloride; Drug: Albuterol Sulfate HFA 0.18 mg (Reference)
- Test 0.09 mg (Experimental)
  Interventions: Other: Methacholine Chloride; Drug: Albuterol Sulfate HFA 0.09 mg (Test)
- Test 0.18 mg (Experimental)
  Interventions: Other: Methacholine Chloride; Drug: Albuterol Sulfate HFA 0.18 mg (Test)

INTERVENTIONS:
Other: Methacholine Chloride — Serial Methacholine dilutions
Drug: Albuterol Sulfate HFA 0.09 mg (Reference) — One actuation each from the Reference inhalation aerosol and the placebo Reference inhalation aerosol and one actuation each from two different placebo Test inhalation aerosols.
  Other Names: Reference single dose
  Arms: Reference 0.09 mg
Drug: Albuterol Sulfate HFA 0.18 mg (Reference) — One actuation each from two different Reference inhalation aerosols and one actuation each from two different placebo Test inhalation aerosols.
  Other Names: Reference double dose
  Arms: Reference 0.18 mg
Drug: Albuterol Sulfate HFA 0.09 mg (Test) — One actuation each from the Test inhalation aerosol and the placebo Test inhalation aerosol and one actuation each from two different placebo Reference inhalation aerosols.
  Other Names: Test single dose
  Arms: Test 0.09 mg
Drug: Albuterol Sulfate HFA 0.18 mg (Test) — One actuation each from two different Test inhalation aerosols and one actuation each from two different placebo Reference inhalation aerosols.
  Other Names: Test double dose
  Arms: Test 0.18 mg
Drug: Placebo — One actuation each from two different placebo Reference inhalation aerosols and one actuation each from two different placebo Test inhalation aerosols.
  Other Names: Test and Ref Placebos
  Arms: Zero dose:

SUMMARY:
Pharmacodynamic bioequivalence study of Albuterol Sulfate Inhalation Aerosol 0.09 mg

DETAILED DESCRIPTION:
To assess the pharmacodynamic bioequivalence of Albuterol Sulfate Inhalation Aerosol 0.09 mg base/ INH [Aurobindo Pharma, USA, Inc] compared to authorized generic drug Albuterol Sulfate HFA Inhalation Aerosol 0.09 mg per actuation [Teva Pharmaceuticals USA, Inc] in stable mild asthma patients, under Methacholine induced bronchoprovocation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female subjects (18-65 years of age).
2. Stable mild asthmatics based on National Asthma Education and Prevention Program (NAEPP) guidelines.
3. FEV1 ≥ 80% of predicted.
4. Airway responsiveness to methacholine demonstrated by a pre-albuterol dose (baseline) PC20 ≤ 8 mg/mL or equivalent PD20.
5. Nonsmokers for at least six months prior to the study and a maximum smoking history of five pack-years (the equivalent of one pack per day for five years).
6. Written informed consent.

Exclusion Criteria:

1. Evidence of upper or lower respiratory tract infection (e.g., pneumonia, bronchitis, sinusitis) within six weeks prior to the study.
2. History of seasonal asthma exacerbations, in which case the subject should be studied outside of the relevant allergen season.
3. History of cystic fibrosis, bronchiectasis or other respiratory diseases.
4. History of cardiovascular, renal, neurologic, liver or endocrine dysfunction, including ECG with evidence of ischemic heart disease.
5. Treatment in an emergency room or hospitalization for acute asthmatic symptoms or need for daily oral corticosteroids within past three months.
6. Known intolerance or hypersensitivity to any component of the albuterol MDI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Post-dose PD20 | Over a period of 4 weeks
  Provocative dose of the methacholine challenge agent required to reduce the forced expiratory volume in one second (FEV1) by 20% following administration of differing doses of albuterol (or placebo) by inhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Marialouis, MD, Study Director — Aurobindo Pharma Ltd
Locations (1):
- Investigational site #1, San Jose, California, United States